CLINICAL TRIAL: NCT04028934
Title: Study of the Quality of Life of Patients Treated by Heavy Surgery as Part of an Enhanced Recovery at Beau Soleil Clinic- QUALICHIR
Acronym: QUALICHIR
Status: Completed | Type: Observational
Sponsor: Clinique Beau Soleil (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A01140-55
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Enhanced Recovery After Surgery; Cystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heavy and oncological surgery is undergoing a major evolution. Some surgical dogmas are falling and care is better rationalized. The interactions between the patient and the caregivers on the other hand, and from the caregiver to the caregiver are favored. Thus was born, about 10 years ago, the principle of enhanced recovery after surgery (ERAS).

But recovery has improved in the patient in the best possible shape in the operating room, and, during the gesture, minimize the negative effects of surgery and anesthesia. Finally, postoperatively, to re-empower the patient as quickly as possible.

The interest of this study is the benefit of the quality of life of the patient being treated for cystectomy as part of an enhanced recovery program. This is to argue the diffusion of this program and the care teams for its realization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication of cystectomy validated by the surgical team and if there is an oncological indication by the multidisciplinary meeting of onco-urology.
* Patient affiliated to a social security scheme
* Patient classified ASA from 1 to 3
* Patient informed and having accepted the principle of enhanced recovery after surgery

Exclusion Criteria:

* Patients classified ASA ≥4
* Patients with severe or poorly balanced associated conditions (diabetes, long-term corticosteroid therapy, severe undernutrition, cirrhosis, immunosuppression, cardiac disease), contraindications to enhanced recovery after surgery (ERAS) may be temporary if they are corrected.
* Patients who can not comply with the ERAS protocol because they do not understand the language or cognitive disorder.
* Vulnerable people (Article L 1121-6 of the CSP)
* Majors subject to legal protection or unable to express their consent (Article 1121-8 of the CSP)

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with an indication of cystectomy validated by the surgical team and if there is an oncological indication by the multidisciplinary meeting of onco-urology, and having accepted the principle of ERAS
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Estimation of the percentage of patients who will have a "good or very good" quality of life, when they were included in an enhanced recovery program in urology following a cystectomy | 6 months
  An overall quality of life questionnaire adapted to each pathology, on a five-level Likert scale, will make it possible to estimate the percentage of patients whose quality of life will be "good or very good".
  The quality of life will be estimated globally through repeated measurements at each visit. It will be considered that if more than 80% of the answers are "good or very good", the quality of life variable will be "good or very good".

CONTACTS AND LOCATIONS:
Locations (1):
- Lacombe Sandy, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided